CLINICAL TRIAL: NCT01110330
Title: A Double-Blind, Randomized, Parallel Group Comparison of Nizoral Cream (F012), Ketoconazole 2% Cream (F126) and Placebo (F000) in the Treatment of Interdigital Tinea Pedis
Brief Title: An Efficacy Study of a New Formulation of Ketoconazole 2% Cream in Patients With Tinea Pedis, Commonly Known as Athlete's Foot
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unexpected discordant results between the KOH microscopy and mycological culture tests at three study sites in the UK.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR012910; KETFUN3001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Tinea Pedis
Keywords: Tinea Pedis; Ketoconazole (NIZORAL); Antifungal Agents; Miconazole (DAKTARIN)
MeSH Terms: conditions — Tinea Pedis | interventions — Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketoconazole 2% cream (formulation F126) (Experimental): ketoconazole 2% cream (formulation F126) A topical white homogenous cream containing the equivalent of 20 mg (or 2%) of ketoconazole applied sparingly to all affected areas of the foot (or feet) once daily (at night or in the evenings) for a total of 4 weeks.
  Interventions: Drug: Ketoconazole 2% cream (formulation F126)
- Ketoconazole 2% cream (formulation F012) (Nizoral) (Experimental): ketoconazole 2% cream (formulation F012) (Nizoral) A topical white homogenous cream containing the equivalent of 20 mg (or 2%) of ketoconazole identical in appearance to study drug applied sparingly to all affected areas of the foot (or feet) once daily (at night or in the evenings) for a total of 4 weeks.
  Interventions: Drug: Ketoconazole 2% cream (formulation F012) (Nizoral)
- Placebo cream (Placebo Comparator): Placebo cream A topical white homogenous cream identical in appearance to study drug applied sparingly to all affected areas of the foot (or feet) once daily (at night or in the evenings) for a total of 4 weeks.
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: Placebo cream — A topical, white, homogenous cream identical in appearance to study drug applied sparingly to all affected areas of the foot (or feet), once daily (at night or in the evenings) for a total of 4 weeks.
  Arms: Placebo cream
Drug: Ketoconazole 2% cream (formulation F012) (Nizoral) — A topical, white, homogenous cream containing the equivalent of 20 mg (or 2%) of ketoconazole identical in appearance to study drug applied sparingly to all affected areas of the foot (or feet), once daily (at night or in the evenings) for a total of 4 weeks.
  Arms: Ketoconazole 2% cream (formulation F012) (Nizoral)
Drug: Ketoconazole 2% cream (formulation F126) — A topical, white, homogenous cream containing the equivalent of 20 mg (or 2%) of ketoconazole applied sparingly to all affected areas of the foot (or feet), once daily (at night or in the evenings) for a total of 4 weeks.
  Arms: Ketoconazole 2% cream (formulation F126)

SUMMARY:
The purpose of this study is to determine if a new formulation of ketoconazole 2% cream is as effective as a current formulation of ketoconazole 2% cream (Nizoral) compared with placebo in treating patients with Tinea pedis, a skin infection commonly known as "athlete's foot" that is caused by a kind of mold called a fungus.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither the physician nor the patient knows the name of the assigned treatment), multicentre study in Poland and the United Kingdom designed to assess the mycological (fungal) cure rate and clinical efficacy of a new formulation of ketoconazole 2% cream (F126) with the current formulation of ketoconazole 2% cream (Nizoral) (F012) compared with placebo cream in patients with symptomatic uncomplicated interdigital (between the toes) Tinea pedis, a skin infection commonly known as "athlete's foot" that is caused by a kind of mold called a fungus. Approximately 548 patients who have symptomatic uncomplicated interdigital Tinea pedis confirmed by positive potassium hydroxide (KOH) microscopy (examination using a microscope) and mycological (fungal) culture will be randomized to receive 1 of 2 formulations of ketoconazole 2% cream (formulation F012 or F126) or placebo cream. There will be 4 study visits during the study. At Visit 1 (baseline), patients will sign the informed consent and be assessed for mycological and clinical signs and symptoms of Tinea pedis. Baseline demographics (age, race, etc), medical history and medication (s) that the patient is currently taking will be recorded. Patients will be issued with a tube of the cream and instructed to apply the cream sparingly to all affected areas of the foot (or feet), once daily (at night or in the evenings) for a total of 4 weeks according to protocol-specified guidelines. During the 4-week treatment period patients will return to the study every 2 weeks to be assessed for clinical signs and symptoms. After the 4-week treatment period, patients will continue participation in the study for an additional 2 weeks without medication. Patients will return then return to the study center for a final visit (Visit 4, Week 6) at which time skin scrapings will be sampled from interdigital spaces on both feet for KOH microscopy and mycological culture. The primary efficacy endpoint is to determine whether a new formulation of ketoconazole 2% cream is equivalent (or as effective) as the current formulation of ketoconazole 2% cream (Nizoral) compared to a placebo cream in achieving a mycological cure (defined as negative KOH microscopy and negative mycological culture) following 4 weeks of treatment. The primary outcome measure in the study is a mycological cure (defined as negative KOH microscopy and negative mycological culture) at week 6. Patients will be monitored for safety (occurrence of adverse events, use of concomitant medications, and reasons for premature discontinuation from the study) from Visit 1 through Visit 4 (Week 6 or time of early termination from study). Patients will be provided with up to two 15g tubes of ketoconazole cream (formulation F126 or F012) or matching placebo cream and be instructed to apply cream sparingly to affected areas of the feet once daily at night or in the evening for 4 weeks according to protocol specified guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Be co-operative, reliable and sufficiently competent to grade and record symptoms as requested
* have a clinical diagnosis of uncomplicated interdigital Tinea pedis confirmed by KOH microscopy
* Be either post-menopausal or surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control before entry and throughout the study and have a negative urine pregnancy test at screening (applies to women only)
* Sign an informed consent form indicating an understanding of the purpose of and procedures required for the study and willingness to participate in the study

Exclusion Criteria:

* Have complicated Tinea pedis defined as confluent, diffuse moccasin type tinea pedis of the entire plantar surface (undersurface of foot), onychomycosis (fungal nail infection)
* other dermatomycosis (fungal skin infection) requiring active treatment
* Have a previous sensitivity to imidazole antifungal agents or to any ingredient of the study medication
* Have a history of disallowed therapies including oral (by mouth) antifungal treatments within the previous 6 weeks, recent use (within 2 weeks of the study start) of topical antifungal agent, immunosuppressive or radiation therapy within the previous 4 weeks, recent use (within 2 weeks prior to screening) of other oral antibiotics, systemic corticosteroids or topical corticosteroids or antibiotics applied to the feet
* Be HIV-positive (testing will not be performed)
* Have uncontrolled diabetes mellitus or peripheral vascular disease requiring active treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (11):
- Poland (4):
  - Bydgoszcz
  - Lodz
  - Lublin
  - Torun
- United Kingdom (7):
  - Cardiff
  - Chorley
  - Glasgow
  - Liverpool
  - Manchester
  - Reading
  - Sunbury-on-Thames

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All randomized patients (583) received at least one dose of study treatment and were included in the Safety Set. Only patients who had a positive Tinea pedis culture at baseline, ie 281 patients, were included in the Positive Baseline Culture Set (PBCS), which was the set used for analysis of the Primary and Secondary Outcome Measures.
Groups:
- Placebo: A topical white homogenous cream identical in appearance to study drug
- Nizoral: Ketoconazole 2% cream (formulation F012) (Nizoral)
- Ketoconazole: Ketoconazole 2% cream (formulation F126)
Period: Overall Study
Arm/Group | Placebo | Nizoral | Ketoconazole
Started | 119 | 230 | 234
Positive Baseline Culture Set | 56 | 111 | 114
Completed | 104 | 207 | 208
Not Completed | 15 | 23 | 26
Not completed — Adverse Event | 0 | 4 | 3
Not completed — Lack of Efficacy | 3 | 1 | 1
Not completed — Lost to Follow-up | 9 | 10 | 15
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 6 | 2
Not completed — Other | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nizoral | Ketoconazole | Total
Number analyzed (Participants) | 119 | 230 | 234 | 583
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 0 | 3
  Between 18 and 65 years | 109 | 207 | 209 | 525
  >=65 years | 9 | 21 | 25 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (14.89) | 45 (13.94) | 45.9 (14.62) | 45 (14.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 71 | 61 | 161
  Male | 90 | 159 | 173 | 422
Baseline BMI [Mean (Standard Deviation); unit: kg/m2] | 28.1 (5.81) | 27.9 (4.76) | 28.3 (5.09) | 28.1 (5.11)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients in the Positive Baseline Culture Set (PBCS) With Mycological Cure (MC) at Week 6
Description: Mycological Cure (MC) was defined as having a negative potassium hydroxide (KOH) microscopy and negative fungal culture at Week 6.
Time Frame: Week 6
Population: Only patients who had a positive Tinea pedis culture at baseline, ie 281 patients, were included in the Positive Baseline Culture Set (PBCS), which was the set used for analysis of the Primary Outcome Measure.
Measure: Number; unit: participants
Arm/Group | Placebo | Nizoral | Ketoconazole
Number analyzed (Participants) | 56 | 111 | 114
participants | 11 | 64 | 64

2. Secondary Outcome: The Number of Patients in the Positive Baseline Culture Set (PBCS) With Overall Cure (OC) at Week 6
Description: Overall Cure (OC) was defined as Mycological Cure (MC) in addition to a global clinical evaluation of either 'Completely Cleared' (clearance of all signs and symptoms of Tinea pedis) or 'Marked Improvement' (significant improvement of signs and symptoms of Tinea pedis; residual signs and symptoms only), assessed at Week 6.
Time Frame: Week 6
Population: Only patients who had a positive Tinea pedis culture at baseline, ie 281 patients, were included in the Positive Baseline Culture Set (PBCS), which was the set used for analysis of the Secondary Outcome Measure.
Measure: Number; unit: participants
Arm/Group | Placebo | Nizoral | Ketoconazole
Number analyzed (Participants) | 56 | 111 | 114
participants | 5 | 55 | 50

ADVERSE EVENTS:
Arm/Group | Ketoconazole | Nizoral | Placebo
Serious Adverse Events (participants affected / at risk) | 2/234 | 5/230 | 2/119
Other Adverse Events (participants affected / at risk) | 55/234 | 50/230 | 28/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketoconazole (N=234) | Nizoral (N=230) | Placebo (N=119)
Anal Abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Benign Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1
Renal Colic (Renal and urinary disorders) | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ketoconazole (N=234) | Nizoral (N=230) | Placebo (N=119)
Palpitations (Cardiac disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Loose Tooth (Gastrointestinal disorders) | 1 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Application Site Erythema (General disorders) | 0 | 0 | 1
Application Site Pruritus (General disorders) | 0 | 1 | 0
Application Site Reaction (General disorders) | 1 | 1 | 0
Chest Discomfort (General disorders) | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 1
Oedema Peripheral (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 2 | 0
Nasopharyngitis (Infections and infestations) | 6 | 3 | 3
Oral Candidiasis (Infections and infestations) | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 1 | 0
Rhinitis (Infections and infestations) | 2 | 2 | 0
Tinea Pedis (Infections and infestations) | 3 | 5 | 6
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth Infection (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 2 | 5
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 0
Wound Infection (Infections and infestations) | 0 | 1 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Human Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Muscle Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Procedural Nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skeletal Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Biopsy (Investigations) | 0 | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 1 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 2
Lethargy (Nervous system disorders) | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Tooth Extraction (Surgical and medical procedures) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated prematurely by the sponsor due to significant discrepancies between potassium hydroxide and mycological culture results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No